CLINICAL TRIAL: NCT03812497
Title: Interplay Between Pediatric Obesity Related Plasma Metabolite Profile and Gut Microbiota
Brief Title: Pediatric Obesity Related Metabolite Profile and Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ky Young Cho, Associate professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Microbiome and metabolome
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Obesity, Childhood
Keywords: Microbiome; Metabolome
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Intervention arm: every obese children will have individualized education program about diet control and exercise in usual life.
  Control arm: normal weight children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese Children Group (Experimental): To reduce the weight, every obese children will receive individualized education program about a way of dietary control and exercise in their usual life. This individualized education program, developed by investigators, specialized dietitian and exercise teacher, is scheduled once a month.
  Interventions: Behavioral: Individualized Education Program
- Normal Weight Children Group (No Intervention): Normal weight children

INTERVENTIONS:
Behavioral: Individualized Education Program — The every participants will have individualized education program about a way of dietary control and exercise in their usual life.
  Arms: Obese Children Group

SUMMARY:
In this study, the investigators aimed to observe changes in the gut microbial composition before and after the weight-loss intervention, including dietary control and exercise, in obese children. The main metabolites produced by gut microbiome, short chain fatty acids (SCFAs) will be also analysed. The investigators will analyse the change of gut microbiome composition and metabolites related with weight-loss intervention and the relationship between microbiome composition and metabolites.

DETAILED DESCRIPTION:
Many recent studies have suggested that dysbiosis of the gut microbiome might related to obesity. There is growing evidence that the composition of gut microbiome changes in childhood obesity compared to normal-weight children, and it is attracting attention as an adjustable environmental factor in obesity treatment. It has been reported that gut microbiome could be changed due to environmental influences such as diet and exercise. In this study, the investigators aimed to observe changes in the gut microbial composition before and after the weight-loss intervention, including dietary control and exercise, in obese children. The main metabolites produced by gut microbiome, short chain fatty acids (SCFAs) would be also analysed to investigate the relationship with gut microbiome and with weight-loss intervention. Intervention is not performed for normal-weight children, and samples from normal-weight children will be used as a control for gut microbiome and biochemical tests.

ELIGIBILITY:
Inclusion Criteria:

* Obese children: Children ≥95 ‰
* Non-obese children: 5‰<BMI <85 ‰

Exclusion Criteria:

* Taking antibiotics, probiotics, or steroids for a month before visit
* Taking probiotics-like products including yogurt for seven days before visit
* Having enteritis symptoms including diarrhea for a month before visit
* Chronic heart disease, chronic bowel disease, chronic liver disease, chronic kidney disease, endocrine disease, genetic diseases or congenital metabolic disorder

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2021-06-28 (Estimated); Study Completion 2021-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiome composition in stool samples | up to 3 months after enrollment
  Bacterial diversity and composition using 16s rRNA sequencing. Especially Bacteroidetes and Firmicutes populations in fecal microbiome will be analyzed related with obesity.

SECONDARY OUTCOMES:
Changes in short chain fatty acids of fecal samples | up to 12 months after enrollment
  The main metabolites produced by gut microbiome, short chain fatty acids using gas chromatography- mass-spectrometry.

OTHER OUTCOMES:
The relationship between gut microbiome composition and fecal short chain fatty acid | up to 12 months after enrollment
  The relationship between gut microbiome composition and metabolites will be analyzed by canonical correspondence analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ky Young Cho, Ph.D., Principal Investigator — Kangnam Sacred Heart Hospital, Hallym University College of Medicine
Locations (1):
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Study participants will only agree if IPD is not shared.

REFERENCES:
- [Derived] Cho KY. Lifestyle modifications result in alterations in the gut microbiota in obese children. BMC Microbiol. 2021 Jan 6;21(1):10. doi: 10.1186/s12866-020-02002-3. PMID 33407104